CLINICAL TRIAL: NCT05972148
Title: The Accuracy of Intraoral Scanning and Photogrammetry on the Clinical Fit of Long-span Frameworks
Brief Title: Precision of Complete-arch Digital Implant Impressions With Intraoral Scanning Versus Photogrammetry
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: William Negreiros (Other)
Collaborators: ITI International Team for Implantology, Switzerland (Other)
Responsible Party: Sponsor-Investigator, William Negreiros, Research Associate, Harvard School of Dental Medicine
Organization: Harvard School of Dental Medicine (Other)
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: IRB18-0660
Record Dates: First submitted 2023-07-25; First posted 2023-08-02 (Actual); Last update posted 2023-08-03 (Actual); Status verified 2023-08

CONDITIONS: Edentulous Jaw
Keywords: edentulous/edentulism; CAD-CAM; implantology; prosthetic dentistry; clinical studies/trial; clinical outcomes
MeSH Terms: conditions — Jaw, Edentulous; Mouth, Edentulous

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intraoral Scanning (Active Comparator)
  Interventions: Other: Digital scanning
- Photogrammetry Scanning (Experimental)
  Interventions: Other: Photogrammetry

INTERVENTIONS:
Other: Digital scanning — Five intraoral scans, one for each arch before the insertion of scanbodies, were obtained. The implant locations were then marked, and the software trimmed a 6mm diameter circular section of the scan from the implant locations to allow the scanbodies to be added. Abutment-level polyetheretherketone (PEEK) scanbodies were hand-tightened onto each implant and not moved for the remainder of the scans. Scanbodies were scanned using a circular scan path, and scanning was finalized.
  Arms: Intraoral Scanning
Other: Photogrammetry — Rectangular-shaped titanium photogrammetry scanbodies were hand-tightened onto the Implants. Scanbodies were not moved before completing all scans for each arch. A total of five scans of each arch were obtained using a photogrammetry device. Measurements were successfully recorded by turning them green on the computer screen.
  Arms: Photogrammetry Scanning

SUMMARY:
The goal of this cross-over clinical trial is to investigate the precision of digital implant impressions using an intraoral scanner and photogrammetry in obtaining complete-arch implant-supported scans.

The main question[s] it aims to answer are:

* Is there a difference in precision between intraoral scans and photogrammetry in obtaining digital implant scans?
* Will arch perimeter and jaw type (maxilla vs. mandible) affect the precision results?

Procedures: At each appointment, participants existing permanent/temporary prosthesis or healing caps were unscrewed and temporarily removed for the period of the consultation appointment.

Scanbodies were screwed into their implants for the duration of the appointment.

They underwent two types of digital implant impression procedures (five times each), including intraoral scan and photogrammetry.

Intraoral and extraoral photography were taken.

At the end of each appointment, the scanbodies were removed, and existing bridge/healing caps were reinserted.

The procedures were not painful or required any form of local anesthetic

Comparison group: Researchers compared the precision of intraoral scanning vs. photogrammetry to see which device provided the best precision outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Present with a completely edentulous arch with at least four implants
* Have bone-level implants
* Intended for restoration with a screw-retained abutment-level fixed implant-supported prosthesis.

Exclusion Criteria:

* Patients unable to tolerate the digital scans impressions
* Presented with implants other than bone-level platforms
* Not intended for restorations with screw-retained abutment-level fixed implant-supported prosthesis
* Not completely edentulous.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2019-08-12 (Actual); Primary Completion 2020-09-20 (Actual); Study Completion 2022-05-02 (Actual)

PRIMARY OUTCOMES:
To investigate the precision of intraoral scanner compared with photogrammetry in performing complete-arch digital implant impressions | During procedure [two hours]

CONTACTS AND LOCATIONS:
Overall Officials: German O Gallucci, DMD, Study Chair — Harvard School of Dental Medicine
Locations (1):
- Harvard School of Dental Medicine, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No
There are no plans for IPD sharing because the study is complete.